CLINICAL TRIAL: NCT01709071
Title: Double Blind Dose - Escalation, Randomized, Controlled, Phase I-II Trial to Evaluate Safety and Immunogenicity of Three Doses of Sabin-IPV and Adjuvanted Sabin-IPV in Healthy Infants
Brief Title: Safety and Immunogenicity of a New Inactivated Poliovirus Vaccine in Infants
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pauline Verdijk (Other Government)
Collaborators: World Health Organization (Other)
Responsible Party: Sponsor-Investigator, Pauline Verdijk, Clinical Research Scientist, National Institute for Public Health and the Environment (RIVM)
Organization: National Institute for Public Health and the Environment (RIVM) (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NVI-256B; 2011-003792-11 (EudraCT Number)
Record Dates: First submitted 2012-10-16; First posted 2012-10-17 (Estimated); Last update posted 2014-02-21 (Estimated); Status verified 2014-02

CONDITIONS: Poliomyelitis
Keywords: Vaccination; Inactivated poliomyelitis vaccine; poliomyelitis; Sabin strains
MeSH Terms: conditions — Poliomyelitis | interventions — Poliovirus Vaccine, Inactivated

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Low dose Sabin-IPV (Experimental): Intramuscular injection of 0.5 ml of Inactivated Poliomyelitis Vaccine containing 5, 8, 16 D-antigen units respectively of Sabin-1,-2 and -3 per dose.
  Infants receive three vaccinations with an interval of 8 weeks between doses.
  Interventions: Drug: Low dose Sabin-IPV
- Low dose adjuvanted Sabin-IPV (Experimental): Intramuscular injection of 0.5 ml of Inactivated Poliomyelitis Vaccine containing 2.5, 4, 8 D-antigen units respectively of Sabin-1,-2 and -3 per dose adjuvanted with 0.5 mg aluminium hydroxide.
  Infants receive three vaccinations with an interval of 8 weeks between doses.
  Interventions: Drug: Low dose adjuvanted Sabin-IPV
- Middle dose Sabin-IPV (Experimental): Intramuscular injection of 0.5 ml of Inactivated Poliomyelitis Vaccine containing 10, 16, 32 D-antigen units respectively of Sabin-1,-2 and -3 per dose.
  Infants receive three vaccinations with an interval of 8 weeks between doses.
  Interventions: Drug: Middle dose Sabin-IPV
- Middle dose adjuvanted Sabin-IPV (Experimental): Intramuscular injection of 0.5 ml of Inactivated Poliomyelitis Vaccine containing 5, 8, 16 D-antigen units respectively of Sabin-1,-2 and -3 per dose adjuvanted with 0.5 mg aluminium hydroxide.
  Infants receive three vaccinations with an interval of 8 weeks between doses.
  Interventions: Drug: Middle dose adjuvanted Sabin-IPV
- High dose Sabin-IPV (Experimental): Intramuscular injection of 0.5 ml of Inactivated Poliomyelitis Vaccine containing 20, 32, 64 D-antigen units respectively of Sabin-1,-2 and -3 per dose.
  Infants receive three vaccinations with an interval of 8 weeks between doses.
  Interventions: Drug: High dose Sabin-IPV
- High dose adjuvanted Sabin-IPV (Experimental): Intramuscular injection of 0.5 ml of Inactivated Poliomyelitis Vaccine containing 10, 16, 32 D-antigen units respectively of Sabin-1,-2 and -3 per dose adjuvanted with 0.5 mg aluminium hydroxide.
  Infants receive three vaccinations with an interval of 8 weeks between doses.
  Interventions: Drug: High dose adjuvanted Sabin-IPV
- Conventional IPV (Active Comparator): Intramuscular injection of 0.5 ml of Inactivated Poliomyelitis Vaccine containing 40, 8, and 32 D-antigen units respectively of Mahoney, MEF-1 and Saukett poliovirus per dose.
  Infants receive three injections with an interval of 8 weeks between doses.
  Interventions: Drug: IPV

INTERVENTIONS:
Drug: IPV
  Other Names: IPV (NVI); Inactivated poliomyelitis vaccine; Inactivated poliovirus vaccine; Inactivated polio vaccine
  Arms: Conventional IPV
Drug: Low dose Sabin-IPV
  Arms: Low dose Sabin-IPV
Drug: Low dose adjuvanted Sabin-IPV
  Arms: Low dose adjuvanted Sabin-IPV
Drug: Middle dose Sabin-IPV
  Arms: Middle dose Sabin-IPV
Drug: Middle dose adjuvanted Sabin-IPV
  Arms: Middle dose adjuvanted Sabin-IPV
Drug: High dose Sabin-IPV
  Arms: High dose Sabin-IPV
Drug: High dose adjuvanted Sabin-IPV
  Arms: High dose adjuvanted Sabin-IPV

SUMMARY:
A new inactivated polio vaccine based on attenuated poliovirus strains was developed to transfer the technology to manufacturers in low- and middle-income countries. This vaccine was produced in different dosages and in different formulations. In healthy adults the safety of the highest dose was comparable to that of the existing inactivated polio vaccine. The purpose of this trial is to determine the safety of the different dosages and formulations of the vaccine in infants. The second goal of this study is to analyse the immune response after three doses in infants.

DETAILED DESCRIPTION:
The goal of this study is to assess the safety and immunogenicity of Sabin-IPV and adjuvanted Sabin-IPV produced with the production process set up for technology transfer by the National Institute for Public Health and the Environment (RIVM, formerly the Netherlands Vaccine Institute (NVI).

* The primary objective is to evaluate safety (local and systemic reactions) of intramuscular injection with Sabin-IPV and adjuvanted Sabin-IPV in healthy infants.
* The secondary objective is to evaluate immunogenicity of three doses Sabin-IPV and adjuvanted Sabin-IPV in infants.

ELIGIBILITY:
Inclusion Criteria:

* Age 8 weeks (56-63 days) at the time of first vaccination
* Infants in good general health, eligible to be vaccinated according to the Polish national vaccination program. The same health criteria apply as used in well-baby clinics when a child receives a vaccination, e.g. also children with a small increase in temperature (< 38.5° C) or with a common cold (runny nose etc) are seen as children with normal health.
* The parent(s)/legally representative(s) have to be willing and able to allow their child to participate in the trial according to the described procedures
* Presence of a signed informed consent in which the parent(s)/legally representative(s) have given written informed consent after receiving oral and written information (signature from one parent in case of single-parent family).

Exclusion Criteria:

* Any IPV or OPV dose
* Known or suspected allergy against any of the vaccine components
* History of unusual or severe reactions to any previous vaccination administration of plasma (including immunoglobulins) or blood products prior and during the study
* Any vaccination less than 14 days before or after each vaccination with the IMP
* History of any neurological disorder including epilepsy or febrile seizures
* Any infectious disease at the time of screening and/or inclusion that might interfere with the results of the study
* Present evidence of serious disease(s) demanding immunosuppressive medical treatment, like cytostatics and prednisolones, that might interfere with the results of the study
* Any known or suspected primary or secondary immunodeficiency
* Communication problems interfering in the study realization according to the judgment of the investigator
* Bleeding disorders and use of anticoagulants
* Premature birth (<37 weeks)
* Participation in another clinical trial

Ages: 56 Days to 63 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2012-02; Primary Completion 2012-11 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Number of adverse reactions following vaccination | 5 days or until adverse reactions have resolved

SECONDARY OUTCOMES:
Level of virus neutralizing titers in serum | 28 days after last vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Verdijk, PhD, Study Director — National Institute for Public Health and the Environment (RIVM)
Locations (7):
- Poland (7):
  - NZOZ Centrum Zdrowia "Błonie", Bydgoszcz
  - Specjalistyczna Poradnia Medyczna "Przylądek Zdrowia", Krakow
  - Szpital im. Jana Pawła II, Krakow
  - Samodzielny Publiczny ZOZ, Lubartów
  - NZOZ Praktyka Lekarza Rodzinnego "Eskulap", Lublin
  - NZLA Michałkowice Jarosz i Partnerzy Spółka Lekarsk, Siemianowice Śląskie
  - Alergo-Med Specjalistyczna Przychodnia Lekarska Sp z o.o., Tarnów

REFERENCES:
- [Background] Bakker WA, Thomassen YE, van't Oever AG, Westdijk J, van Oijen MG, Sundermann LC, van't Veld P, Sleeman E, van Nimwegen FW, Hamidi A, Kersten GF, van den Heuvel N, Hendriks JT, van der Pol LA. Inactivated polio vaccine development for technology transfer using attenuated Sabin poliovirus strains to shift from Salk-IPV to Sabin-IPV. Vaccine. 2011 Sep 22;29(41):7188-96. doi: 10.1016/j.vaccine.2011.05.079. Epub 2011 Jun 7. PMID 21651934
- [Background] Verdijk P, Rots NY, Bakker WA. Clinical development of a novel inactivated poliomyelitis vaccine based on attenuated Sabin poliovirus strains. Expert Rev Vaccines. 2011 May;10(5):635-44. doi: 10.1586/erv.11.51. PMID 21604984
- [Background] Verdijk P, Rots NY, van Oijen MG, Oberste MS, Boog CJ, Okayasu H, Sutter RW, Bakker WA. Safety and immunogenicity of inactivated poliovirus vaccine based on Sabin strains with and without aluminum hydroxide: a phase I trial in healthy adults. Vaccine. 2013 Nov 12;31(47):5531-6. doi: 10.1016/j.vaccine.2013.09.021. Epub 2013 Sep 21. PMID 24063976
- [Derived] Verdijk P, Rots NY, van Oijen MG, Weldon WC, Oberste MS, Okayasu H, Sutter RW, Bakker WA. Safety and immunogenicity of a primary series of Sabin-IPV with and without aluminum hydroxide in infants. Vaccine. 2014 Sep 3;32(39):4938-44. doi: 10.1016/j.vaccine.2014.07.029. Epub 2014 Jul 18. PMID 25043278